CLINICAL TRIAL: NCT01040325
Title: A Phase Two, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of the Travelers' Diarrhea Vaccine System in Travelers to Asia
Brief Title: Traveler's Diarrhea (TD) Vaccine Asia Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ELT209; EudraCT Number: 2009-015603-10
Record Dates: First submitted 2009-12-25; First posted 2009-12-29 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-01

CONDITIONS: Traveler's Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): 358 subjects receive a two vaccination regimen with an LT patch
  Interventions: Biological: TD Vaccine System
- Placebo (Placebo Comparator): 358 subjects receive a two vaccination regimen with placebo patch
  Interventions: Biological: TD Vaccine System

INTERVENTIONS:
Biological: TD Vaccine System — TD Vaccine System containing heat labile enterotoxin of E. coli (LT)
  Arms: Active
Biological: TD Vaccine System — TD Vaccine System Containing Placebo Product
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of the TD Vaccine System to prevent moderate to severe enterotoxin E.coli (ETEC) disease in travelers to India.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age at date of first vaccination
* Good health as determined by medical history and physical inspection
* Females of child-bearing potential must have a negative pregnancy test prior to first and second vaccination in the country of origin; females of child-bearing potential must agree not to become pregnant throughout the duration of study
* Subjects must have planned travel to DC, within 3 hours traveling distance of approved study site(s), for a minimum duration of stay of 7 days (no maximum stay is specified for inclusion).
* Subject must be able to communicate in English

Exclusion Criteria:

* Abnormalities as determined by the Investigator/clinician during physical inspection;
* Participated in research involving investigational product within 30 days before planned date of first vaccination;
* Ever received LT, ETEC, or cholera vaccine;
* History of diarrhea while traveling in a developing country within the last year;
* Women who are pregnant or breastfeeding;
* Clinically significant underlying enteric, pulmonary, cardiac, liver or renal disease;
* History of Irritable Bowel Syndrome;
* Seizure disorder within the last year;
* Current use of immunosuppressive therapy (excluding inhaled steroids) or immunodeficiency;
* Known or suspected alcohol abuse or illicit drug use within the last year;
* Medical history of HIV, HBV, or HCV;
* An employee of a study site;
* Known allergies to any component of the vaccine, including adhesives;
* Planned use of antibiotics with known activity against gram negative facultative anaerobes;
* Planned use of antacids, antidiarrheals, loperamide, bismuth subsalicylate, diphenoxylate or similar from two weeks prior to randomization through the surveillance phase of the study;
* An employee of Intercell (global) or an immediate family member.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 723 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence of cases with vaccine preventable outcome | within 17 days after arrival in destination country

SECONDARY OUTCOMES:
Incidence of moderate/severe diarrhea | within 17 days after arrival in destination country

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, MD, Principal Investigator — University of Zurich
Locations (12):
- Germany (2):
  - Belinger Centrum Reise & Tropenmedizin, Berlin
  - Tropical Medicine and Bernhard-Nocht Ints, Hamburg
- India (5):
  - Dr. Tito's Health Care and Diagnostic Centre, Goa
  - Prabhugaunker's Clinic, Goa
  - Wellesley Medicentre, Kolkata
  - Pushpawati Singhania Research Institute, New Delhi
  - Samvedna Hospital, Varanasi
- United Kingdom (5):
  - Synexus, Reading, Berkshire
  - Bio-Kinetic Europe Ltd, Belfast, Northern Ireland
  - Synexus Ltd, Chorley
  - Guy's Drug Research Unit, London
  - Hospital for Tropical Diseases, London